# Study:

**Continuous Wireless Monitoring of Vital Signs and Automated Alerts of Postsurgical Patient Deterioration.** 

NCT04640415

Statistical analysis plan

Version 1

#### **Primary Outcome Measure:**

Cumulative duration

Cumulative duration of one or more deviations in vital signs. List of vital signs, and normal limits detailed in protocol, whichever comes first.

Vital signs value deviations are calculated per 24 hours of monitoring time.

[Time Frame: First 5 days from randomization or until discharge]

#### **Secondary Outcome Measures:**

Frequency of sustained deviation alerts

Frequency of each of the sustained deviations in vital signs. List of vital signs, and normal limits detailed in protocol.

Number of alarms are calculated as the number of alarms per 24 hours.

[Time Frame: First 5 days from randomization or until discharge, whichever comes first]

- AE during the first 7 days and the first 30 days
- SAE during the first 7 days and the first 30 days

### **Tertiary Outcome Measures:**

1. Length of hospital stay

Length of hospital stay

[Time Frame: 30 days from randomization and 6 months]

2. Patient related post-admission healthcare expenses

Total patient-related healthcare expenses in patients experiencing adverse clinical outcomes compared to patients without such outcomes and the effect of the study intervention on expenses

[Time Frame: 2 years]

3. Staff response time (intervention group only)

Time from the staff is notified by app, until they respond by selecting 'check on patient' in app Stratified according to time of day

[Time Frame: Up to 5th postoperative day or until discharge, whichever comes first]

### **Outcome analysis:**

- Intention to treat analysis
  - Patient outcomes are analyzed based on the randomization groups.
- Per-protocol analysis
  - o Patients included in the intervention are those with:
    - intervention patients with alerts with at least one registered use of the app in relation to an alert, as indicated if the "attend", "postpone/snooze" or "transfer" buttons have been used.

OF

• intervention patients with no alerts, are also included in the intervention group.

AND

- o at least 12 hours of monitoring with valid data transfer.
- Patients in the control-group are all patients from the control group with at least 12 hours of monitoring.

## Data analysis:

- Vital values: Gaps in vital value data were not imputed.
   Durations will be calculated in minutes per 24 hours (1440 minutes) of monitoring.
- Data will be presented with descriptive statistics.

Categorical data will be tested with Fishers exact test.

Continuous data will be tested with Wilcoxon Mann-Whitney U test.

Time-till-event will be tested with cox-regression.

- For statistical tests and alpha of < 0.05 will be considered statistically significant.

**Table 1: Patient demographics** 

| | Control arm<br>N = 200 | Intervention arm N = 200 |
|---|---|---|
| Age, mean | | |
| Male, no (%) | | |
| ASA class | | |
| 1 | | |
| II | | |
| III | | |
| >IV | | |
| Smoking status | | |
| Never smoked | | |
| Former smoker | | |
| Current smoker | | |
| Pack years for former<br>and current smokers<br>(mean) | | |
| Preexisting conditions, n<br>(%) | | |
| COPD | | |
| Vascular insufficiency | | |
| Chronic arterial hypertension | | |
| Diabetes Mellitus | | |
| Type of surgery | | |
| Abdominal | | |
| Vascular | | |
| Urologic | | |
| Orthopedic | | |

Table 2: Primary outcomes - Cumulative duration of deviating vital values per 24 hours

| | Intention to treat analysis | | |
|---|---|---|---|
| | Control arm<br>N = 200 | Intervention arm<br>N = 200 | p-value |
| Total cumulative | | | |
| Respiratory | | | |
| SpO2 < 92 % | | | |
| SpO2 < 88 % | | | |
| SpO2 < 85 % | | | |
| SpO2 < 80 % | | | |
| RF < 5 min <sup>-1</sup> | | | |
| RF < 11 min <sup>-1</sup> | | | |
| RF > 24 min <sup>-1</sup> | | | |
| RF > 30 min <sup>-1</sup> | | | |
| Circulatory | | | |
| HR < 30 min <sup>-1</sup> | | | |
| HR [30 - 40] min <sup>-1</sup> | | | |
| HR > 110 min <sup>-1</sup> | | | |
| HR > 130 min <sup>-1</sup> | | | |
| SBP < 70 mmHg | | | |
| SBP < 90 mmHg | | | |
| SBP > 180 mmHg | | | |
| SBP > 220 mmHg | | | |

Table 3: Secondary outcomes - Median number of alarms for sustained deviations per 24 hours. For control patients the number is the theoretical number of alarms a system would issue.

| | Control arm<br>N = 200 | Intervention arm N = 200 | p-value |
|---|---|---|---|
| Desaturation | | | |
| SpO2 < 92 % for > 60 min | | | |
| SpO2 < 88 % for > 10min | | | |
| SpO2 < 85 % for > 5 min | | | |
| SpO2 < 80 % for > 1 min | | | |
| Bradypnea | | | |
| RF < 5 min <sup>-1</sup> for > 1 min | | | |
| RF < 11 min <sup>-1</sup> for > 15 min | | | |
| Tachypnea | | | |
| RF > 24 min <sup>-1</sup> for > 15 min | | | |
| RF > 30 min <sup>-1</sup> for > 5 min | | | |
| Bradycardia | | | |
| HR < 30 min <sup>-1</sup> for > 1 min | | | |
| HR [30 - 40] min <sup>-1</sup> for > 5 min | | | |
| Tachycardia | | | |
| HR > 110 min <sup>-1</sup> for > 60 min | | | |
| HR > 130 min <sup>-1</sup> for > 30 min | | | |
| Hypotension | | | |
| SBP < 70 mmHg for > 30 min | | | |
| SBP < 90 mmHg for > 60 min | | | |
| Hypertension | | | |
| SBP > 180 mmHg for > 60 min | | | |
| SBP > 220 mmHg for > 30 min | | | |

**Table 4: Tertiary outcomes** 

| | Intention to treat analysis | | Per protocol analysis | |
|---|---|---|---|---|
| | Control arm<br>N = 200 | Intervention arm N = 200 | Control arm<br>N = 280 | Intervention arm N = 120 |
| Serious Adverse Events at 7 days / n (%) | XX (xx %) | XX (xx %) | XX (xx %) | XX (xx %) |
| Serious Adverse Events at 30 days / n (%) | XX (xx %) | XX (xx %) | XX (xx %) | XX (xx %) |
| Death / n (%) | XX (xx %) | XX (xx %) | XX (xx %) | XX (xx %) |
| Length of stay<br>/ days [IQR] | X [X-XX] | X [X-XX] | X [X-XX] | X [X-XX] |
| Reoperation / n (%) | XX (xx %) | XX (xx %) | XX (xx %) | XX (xx %) |